CLINICAL TRIAL: NCT03883282
Title: Influence of Participation in Randomized Controlled Trials on Cardiovascular Patient's Adherence to Medicines' Intake and regUlar viSits to the docTor
Brief Title: Influence of Participation in Randomized Controlled Trials on adheRence to Medicines' Intake and regUlar viSits to the docTor
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: TRUST
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Adherence, Patient
Keywords: patient adherence, randomized clinical trials
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Patients who have been participated in RCT in the period from 2011 to 2018 (study group)
  Interventions: Other: Not Provided
- control group: - Patients who have never participated in RCT
  Interventions: Other: Not Provided

INTERVENTIONS:
Other: Not Provided — Not Provided

SUMMARY:
A prospective non-interventional single-center study aimed to evaluate the influence of participation in international randomized controlled trials (RCT) of cardiovascular patients on their compliance and adherence to medicines' intake and regular visits to the doctor in comparison with those patients, who had never participated in RCT within the outpatient registry PROFILE (prospective, observational study).

ELIGIBILITY:
Inclusion criterion for study group

• All patients of the outpatient register PROFILE who participated in the international randomized clinical trials from 2011 to 2018, (n≈100).

Inclusion criterion for control group

• Patients of the outpatient register PROFILE, who from 2011 to 2018 were observed in the research center for preventive medicine and never participated in international randomized clinical trials (n≈100).

Exclusion criteria for both groups

* Patients whose life status is defined as "dead"
* Patients who refused to participate in our study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be taken from the outpatient register PROFILE
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Assessment of motives of enrollment in a trial and patient's attitude to RCT based on elaborated questionnaires for both groups | on enrollment
  The specially designed questionnaire for the study group includes 9 questions. Based on the data obtained, we will be able to draw conclusions about the motives for participating in RCTs, the level of trust towards a doctor, and adherence to treatment after the end of the RCT.
  The questionnaire for the control group includes 8 questions with 3 possible answers as well. Based on the data obtained, we will determine the level of patient awareness of RCTs and the willingness to participate in the trial in the future. This questionnaire is exploratory, each question is considered individually, which allows us to make a more detailed analysis of various aspects of our study.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No